CLINICAL TRIAL: NCT03905473
Title: Habitual Physical Activity in Patients With Myasthenia Gravis Assessed by Accelerometry and Questionnaire
Brief Title: Physical Activity and Fatigue in Myasthenia Gravis
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Linda Kahr Andersen, Research Physiotherapist, Phd student, Rigshospitalet, Denmark
Other Study IDs: H-18031231 1
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Myasthenia Gravis
Keywords: Survey; Physical Activity; Fatigue
MeSH Terms: conditions — Myasthenia Gravis; Motor Activity; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Accelerometer measurements — To validate the questionnaires about physical activity, some patients will be wearing an accelerometer for one week. An accelerometer is a little device worn in a belt around the hip, which can measure intensity of the patient's activity level. The accelerometer is worn 24 hours a day for one week and is only removed when bathing.

SUMMARY:
Danish patients with myasthenia gravis are asked to answer a validated and international questionnaire about physical activity. Also background questions about their disease and comorbidity are asked. To validate the data about physical activity from the questionnaires 69 patients are asked to wear an accelerometer for 7 days to measure activity level.

DETAILED DESCRIPTION:
Secure digital mails are sent to around1500 patients qua their civil registration number (CPR number) (each resident of Denmark has a permanent unique civil registration number that is provided at birth or immigration to Denmark). The mail contains a link for the software REDCap (© 2018 Vanderbilt University), recommended by Rigshospitalet. REDcap is a secure web application for building and managing online surveys and databases. Patients are, in REDcap, informed about the project, and if interested, asked to sign the included informed content and answer six validated and translated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Danish resident.
* Alive.
* Minimum age 18 years.
* Registered in the Danish Patient Register with diagnosis code 70.0 (ICD-10) or 733.09 (ICD 8).
* Subscribing E-boks (the Danish system for receiving secure digital emails).

Exclusion Criteria:

* I fulfilling the inclusion criteria, then no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish patients diagnosed with myasthenia gravis.
Sampling Method: Non-Probability Sample
Enrollment: 779 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI-20) | 5 minutes
  MFI-20 is a self-reported questionnaire that measures fatigue severity. It contains 20 items and consists of five fatigue domains: mental fatigue, reduced motivation, reduced activity, physical fatigue and general fatigue. The response options consist of five check boxes ranging from "Yes, that is true" to "No, that is not true". The scores in each domain range from 4 to 20, with higher scores indicating higher levels of fatigue. A total fatigue score for all five domains is not used. MFI-20 has been used in several clinical and healthy populations.

SECONDARY OUTCOMES:
The short International Physical Activity Questionnaire (IPAQ) | 3 minutes
  IPAQ short form is used to measure self-reported time spent on physical activity and sedentary behavior. The questionnaire measures four intensity levels of physical activity from none (sedentary) to strenuous physical activity. Patients are asked to report number of hours and minutes per day on the different activity levels.
Insomnia Severity Index (ISI) | 3 minutes
  ISI measures self-reported sleep quality and disturbances during the previous 2 weeks. The ISI comprises seven items assessing the perceived severity of difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 - 4 from less to more severe. The total score is the sum of each individual item and can range from 0 to 28 (28= most severe).
Myasthenia gravis activity of daily living profile (MG-ADL) | 10 minutes
  Impact on daily living is assessed using the MG-ADL. An eight-question survey of symptoms severity, with each response graded from 0 (normal) to 3 (most severe). Questions include ocular, oropharyngeal, respiratory, and extremity functions. Total MG-ADL score ranges from 0 to 24. MG-ADL is also an indirect measurement of disease severity.
Myasthenia gravis quality of life 15-item score (MG-QoL15) | 3 minutes
  MG -specific quality-of-life instrument is a 15-item questionnaire encompassing physical and psychological domains of MG to assess disease-specific Qol in MG patients. Rating consist of a 5-point scale ranging from 0 ("not at all") to 4 ("very much") as to the degree to which patients agree with the given statement summing up to a total score 0-60 points.

OTHER OUTCOMES:
Gender | 5 seconds
  Are you a woman or a man?
Verification of the MG status. | 5 seconds
  Are you diagnosed with MG? (Yes/no/ maybe - still under examination)
Age | 5 seconds
  How old are you? (unit: years)
Job | 5 seconds
  How is your actually job status? (working fulltime/ working part time, student, retired, out of work, early retiree, sick leave).
Smoking | 5 seconds
  Are you a smoker? (Never, ex-smoker, daily smoker, smoker but not every day, using e-cigarettes, using nicotine products)
Comorbidity | 5 seconds
  Are you suffering from any of these conditions? (depression, any other psychiatric disorder, any auto-immune disease, chronic obstructive pulmonary disease, any cardiac diseases, chronic fatigue, sleep apnoea)
How many years diagnosed with MG? | 5 seconds
  Number of years since diagnosis.
Symptoms of MG? | 5 seconds
  The patient register symptoms according to the Myasthenia Gravis Foundation of American clinical classification.
Treatment for MG? | 5 seconds
  The patient report their pharmacological treatment for MG.
Are you receiving immunoglobulin treatment or plasmaphereses? | 5 seconds
  Answer yes/no.
Have you had a thymectomy? | 5 seconds
  Answer yes/no.
Are you having any of these treatments? | 5 seconds
  The patient answer yes or no to the following treatments: benzodiazepine, antidepressant drugs or betablockers.
Are you reguarly seen by a neurologist? | 5 seconds
  Answer yes/no
How tall are you? | 2 seconds
  Answer in centimeter
How much do you weight? | 2 seconds
  Answer in kilograms
Are you living alone? | 2 seconds
  Yes/no
Do you live with children? How many? | 2 seconds
  Answer in number of children
Was is your highest education level? | 2 seconds
  Short/middle/high education level

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark